CLINICAL TRIAL: NCT06118164
Title: Effect of Pursed-lips Breathing Combined With Aerobic Walking Exercise on Oxygenation and Activity Endurance in Lung Cancer Patients After Lobectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Tzu Chi Hospital (Other)
Responsible Party: Principal Investigator, Jeng-Yuan Wu, Director of Thoracic Surgery, Taichung Tzu Chi Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TaichungTCH
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Complications During Rehabilitation Stay
Keywords: lung cancer; lobectomy; pursed-lip breathing; aerobic walking; oxygenation; exercise tolerance
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: The experimental group was given pursed-mouth breathing training combined with aerobic walking exercise.
  Control group I was given pursed-mouth breathing training. Control group II was given aerobic walking exercise.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients who agreed to participate were randomly assigned to the experimental group or one of the two control groups (Control I and Control II) by outpatient nurses drawing lots from a lottery box. Once the group assignment was determined, on the day of admission, the researchers provided instructions on the respective intervention measures for that group (Pursed-lip breathing combined with aerobic walking exercise group, Pursed-lip breathing only group, Aerobic walking exercise only group). Data collection was carried out by registered nurses with at least two years of clinical experience in non-enrollment wards.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- experimental group -pursing- lip breathing combined with aerobic walking exercise (Experimental): For the pursed-lip breathing combined with aerobic walking exercise group (experimental group), subjects were taught to coordinate their breathing with their walking. They were instructed to inhale for two steps and exhale with pursed lips for four to five steps. Initially, they were allowed to walk at a pace that felt comfortable to them, and then gradually increase their walking speed until they reached the target aerobic heart rate, calculated using the formula: (220 - age) × 55-65% of maximum heart rate.
  During the walking exercise, a pulse oximeter was used to monitor their heart rate and blood oxygen saturation. Training sessions were conducted daily from the first day after surgery until the fifth day, with three sessions each day, and each session lasting for 15 minutes.
  Interventions: Behavioral: pursing- lip breathing combined with aerobic walking exercise
- Control group 1-pursed-lip breathing (Active Comparator): For the group receiving single pursing- lip breathing training (control group 1), subjects were taught to perform deep inhalation through the nose (counting mentally from 1 to 2) while in a seated or standing position. They were then instructed to purse their lips and exhale slowly and steadily (counting mentally from 1 to 4).
  During the walking exercise, a pulse oximeter was used to monitor their heart rate and blood oxygen saturation. Training sessions were conducted daily from the first day after surgery until the fifth day, with three sessions each day, and each session lasting for 15 minutes.
  Interventions: Behavioral: pursing- lip breathing
- Control group 2 -aerobic walking exercise (Active Comparator): For the single aerobic walking exercise group (control group 2), subjects were taught to start with their own acceptable stride and pace and then gradually increase their walking speed until they reached the target aerobic heart rate. Pulse oximeters were used to monitor their heart rate and blood oxygen saturation levels during the process.
  During the walking exercise, a pulse oximeter was used to monitor their heart rate and blood oxygen saturation. Training sessions were conducted daily from the first day after surgery until the fifth day, with three sessions each day, and each session lasting for 15 minutes.
  Interventions: Behavioral: aerobic walking exercise

INTERVENTIONS:
Behavioral: pursing- lip breathing combined with aerobic walking exercise — pursing- lip breathing combined with aerobic walking exercise
  Arms: experimental group -pursing- lip breathing combined with aerobic walking exercise
Behavioral: pursing- lip breathing — pursing- lip breathing
  Arms: Control group 1-pursed-lip breathing
Behavioral: aerobic walking exercise — aerobic walking exercise
  Arms: Control group 2 -aerobic walking exercise

SUMMARY:
The effects of pursed-lip breathing or aerobic walking exercise in increasing muscle strength and motility and relieving dyspnea have been proved. However, patients with lung cancer often have decreased lung function and exercise capacity after lobectomy. The aim of this study was to explore the effects of pursed-lip breathing combined with aerobic walking exercise on postoperative oxygenation and exercise tolerance of lung cancer patients underwent lobectomy.

DETAILED DESCRIPTION:
An randomized controlled trial was used. Sixty eligible subjects from the Department of Thoracic Surgery of a regional hospital in central Taiwan participate in this study. A total of sixty subjects were randomly and equally assigned to the experimental group, control group I and control group II, to carry out postoperative both pursed lip breathing and aerobic walking exercise, pursed lip breathing, and aerobic walking exercise respectively. All three interventions were conducted 3 times a day, each lasting 15 minutes, from the 1st to 5th day after the operation. Pretests were done before the start of the three interventions on the first postoperative day, and posttests were done after the completion of the three interventions on the 5th postoperative day. Data including 6-minute walking test, Dyspnea Visual Analogue Scale, Rating scale of perceived exertion, peak expiratory flow rate and SpO2 were collected.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged over 20 who have been informed of the research process and are willing to participate and sign consent.
* Participants with clear consciousness, the ability to communicate in Mandarin or Taiwanese, and the ability to walk independently.
* Participants diagnosed with lung cancer who have undergone lung lobe resection surgery.

Exclusion Criteria:

* Changes in the surgical plan, not undergoing at least a single lung lobe resection.
* Deterioration of postoperative condition, making it impossible to correctly perform pursed lip breathing or aerobic walking exercises.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Effect on Postoperative Oxygenation in Lung Cancer Patients | pretests(before the start of the three interventions on the post-op day 1)
  Measurements were taken on the 1st day after surgery, prior to the intervention. The pulse oximeter was placed on the patient's fingertip, and after a 5-second wait, the SpO2 value appeared on the monitor interface, which was then recorded on the data sheet.
Effect on Postoperative Oxygenation in Lung Cancer Patients | posttests(after the completion of the three interventions on the post-op day 5)
  Measurements were taken on the 5th day after surgery, after three activities. The pulse oximeter was placed on the patient's fingertip, and after a 5-second wait, the SpO2 value appeared on the monitor interface, which was then recorded on the data sheet.
Effect on Postoperative Oxygenation in Lung Cancer Patients | pretests(before the start of the three interventions on the post-op day 1)
  Dyspnea Visual Analogue Scale (DVAS):Draw a vertical 10 cm line on an A4 white paper. Label the top end of the line as "Not Breathless" and the bottom end as "Very Breathless." The longer the distance marked on the line, the more severe the breathlessness.
  Measurement Method: Measurements were taken on the 1st day after surgery, prior to the intervention. After the patient completes a six-minute walk test, they mark their level of breathlessness on the vertical line to assess the degree of breathlessness.
Effect on Postoperative Oxygenation in Lung Cancer Patients | posttests(after the completion of the three interventions on the post-op day 5)
  Dyspnea Visual Analogue Scale (DVAS): Draw a vertical 10 cm line on an A4 white paper. Label the top end of the line as "Not Breathless" and the bottom end as "Very Breathless." The longer the distance marked on the line, the more severe the breathlessness.
  Measurement Method: Measurements were taken on the 5th day after surgery, after three activities. After the patient completes a six-minute walk test, they mark their level of breathlessness on the vertical line to assess the degree of breathlessness.
Effect on Postoperative activity endurance in Lung Cancer Patients | pretests(before the start of the three interventions on the post-op day 1)
  Six-minute walking test (6MWT) : A long, flat, unobstructed hospital corridor is selected as the testing location. The floor is marked every 1 meter, covering a total distance of 30 meters. Patients are instructed to walk back and forth within the marked distance. Before the test, patients are informed to walk at the fastest pace they can tolerate and that they can slow down or pause if they experience any physical discomfort during the test. The test lasts for six minutes, and when the time is up, patients stop walking. The location where patients stop is recorded, corresponding to a marked point on the floor. The distances covered are summed up to determine the test result.
Effect on Postoperative activity endurance in Lung Cancer Patients | posttests(after the completion of the three interventions on the post-op day 5)
  Six-minute walking test (6MWT) : A long, flat, unobstructed hospital corridor is selected as the testing location. The floor is marked every 1 meter, covering a total distance of 30 meters. Patients are instructed to walk back and forth within the marked distance. Before the test, patients are informed to walk at the fastest pace they can tolerate and that they can slow down or pause if they experience any physical discomfort during the test. The test lasts for six minutes, and when the time is up, patients stop walking. The location where patients stop is recorded, corresponding to a marked point on the floor. The distances covered are summed up to determine the test result. Measurements were taken on the 1st day after surgery before the intervention.
Effect on Postoperative activity endurance in Lung Cancer Patients | pretests(before the start of the three interventions on the post-op day 1)
  Rating scale of perceived exertion (RPE / Borg 6-20):This scale ranges from 6 points (indicating no perceived exertion) to 20 points (indicating maximal exertion). Higher scores indicate a higher level of perceived exertion.Measurements were taken on the 1st day after surgery before the intervention. After the six-minute walking test, patients were asked to circle the score on the scale that corresponds to their perceived level of exertion to assess the level of exertion felt by patients after activity.
Effect on Postoperative activity endurance in Lung Cancer Patients | posttests(after the completion of the three interventions on the post-op day 5)
  Rating scale of perceived exertion (RPE / Borg 6-20):This scale ranges from 6 points (indicating no perceived exertion) to 20 points (indicating maximal exertion). Higher scores indicate a higher level of perceived exertion.Measurements were taken on the 5th day after surgery after three separate activities. Following the six-minute walking test, patients were asked to circle the score on the scale that corresponds to their perceived level of exertion to assess the level of exertion felt by patients after activity.

CONTACTS AND LOCATIONS:
Overall Officials: Hua-Shan Wu, PhD, Principal Investigator — Asia University
Locations (1):
- Asia University, Taichung, Wufeng, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Amin MB, Greene FL, Edge SB, Compton CC, Gershenwald JE, Brookland RK, Meyer L, Gress DM, Byrd DR, Winchester DP. The Eighth Edition AJCC Cancer Staging Manual: Continuing to build a bridge from a population-based to a more "personalized" approach to cancer staging. CA Cancer J Clin. 2017 Mar;67(2):93-99. doi: 10.3322/caac.21388. Epub 2017 Jan 17. PMID 28094848
- [Result] Abbas AE. Surgical Management of Lung Cancer: History, Evolution, and Modern Advances. Curr Oncol Rep. 2018 Nov 13;20(12):98. doi: 10.1007/s11912-018-0741-7. PMID 30421260
- [Result] Ettinger DS, Wood DE, Aggarwal C, Aisner DL, Akerley W, Bauman JR, Bharat A, Bruno DS, Chang JY, Chirieac LR, D'Amico TA, Dilling TJ, Dobelbower M, Gettinger S, Govindan R, Gubens MA, Hennon M, Horn L, Lackner RP, Lanuti M, Leal TA, Lin J, Loo BW Jr, Martins RG, Otterson GA, Patel SP, Reckamp KL, Riely GJ, Schild SE, Shapiro TA, Stevenson J, Swanson SJ, Tauer KW, Yang SC, Gregory K; OCN; Hughes M. NCCN Guidelines Insights: Non-Small Cell Lung Cancer, Version 1.2020. J Natl Compr Canc Netw. 2019 Dec;17(12):1464-1472. doi: 10.6004/jnccn.2019.0059. PMID 31805526
- [Result] Granger CL, Edbrooke L, Denehy L. The nexus of functional exercise capacity with health-related quality of life in lung cancer: how closely are they related? Ann Transl Med. 2018 Dec;6(Suppl 2):S131. doi: 10.21037/atm.2018.12.35. No abstract available. PMID 30740452
- [Result] Kobayashi N, Kobayashi K, Kikuchi S, Goto Y, Ichimura H, Endo K, Sato Y. Long-term pulmonary function after surgery for lung cancer. Interact Cardiovasc Thorac Surg. 2017 May 1;24(5):727-732. doi: 10.1093/icvts/ivw414. PMID 28453808
- [Result] Lugg ST, Agostini PJ, Tikka T, Kerr A, Adams K, Bishay E, Kalkat MS, Steyn RS, Rajesh PB, Thickett DR, Naidu B. Long-term impact of developing a postoperative pulmonary complication after lung surgery. Thorax. 2016 Feb;71(2):171-6. doi: 10.1136/thoraxjnl-2015-207697. PMID 26769017
- [Result] Li J, Guo NN, Jin HR, Yu H, Wang P, Xu GG. Effects of exercise training on patients with lung cancer who underwent lung resection: a meta-analysis. World J Surg Oncol. 2017 Aug 23;15(1):158. doi: 10.1186/s12957-017-1233-1. PMID 28835249
- [Result] Mayer AF, Karloh M, Dos Santos K, de Araujo CLP, Gulart AA. Effects of acute use of pursed-lips breathing during exercise in patients with COPD: a systematic review and meta-analysis. Physiotherapy. 2018 Mar;104(1):9-17. doi: 10.1016/j.physio.2017.08.007. Epub 2017 Aug 31. PMID 28969859
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Travis WD, Brambilla E, Burke AP, Marx A, Nicholson AG. Introduction to The 2015 World Health Organization Classification of Tumors of the Lung, Pleura, Thymus, and Heart. J Thorac Oncol. 2015 Sep;10(9):1240-1242. doi: 10.1097/JTO.0000000000000663. No abstract available. PMID 26291007
- [Result] Villeneuve PJ. Interventions to avoid pulmonary complications after lung cancer resection. J Thorac Dis. 2018 Nov;10(Suppl 32):S3781-S3788. doi: 10.21037/jtd.2018.09.26. PMID 30505565
- [Result] Ziarnik E, Grogan EL. Postlobectomy Early Complications. Thorac Surg Clin. 2015 Aug;25(3):355-64. doi: 10.1016/j.thorsurg.2015.04.003. Epub 2015 Jun 12. PMID 26210931